CLINICAL TRIAL: NCT06120491
Title: A Randomized, 2-cohort, Double-blind, Placebo-controlled, Phase III Study of Saruparib (AZD5305) in Combination With Physician's Choice New Hormonal Agents in Patients With HRRm and Non-HRRm Metastatic Castration-Sensitive Prostate Cancer (EvoPAR-Prostate01)
Brief Title: Saruparib (AZD5305) vs Placebo in Men With Metastatic Castration-Sensitive Prostate Cancer Receiving Physician's Choice New Hormonal Agents
Acronym: EvoPAR-PR01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9723C00001; 2023-504214-30-00 (Other: EU CTIS)
Record Dates: First submitted 2023-10-17; First posted 2023-11-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-Sensitive Prostate Cancer
Keywords: AZD5305; Saruparib; HRRm; non-HRRm; mCSPC; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — AZD5305; Abiraterone Acetate; darolutamide; enzalutamide

STUDY DESIGN:
Intervention Model Description: within each cohort (HRRm and non-HRRm), participants are randomised in 1:1 ratio to one of two treatment arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Saruparib (AZD5305) + Physician's Choice NHA (Experimental): Saruparib (AZD5305) + physician's choice NHA (Abiraterone, Darolutamide, or Enzalutamide)
  Interventions: Drug: Saruparib; Drug: Abiraterone Acetate; Drug: Darolutamide; Drug: Enzalutamide
- Arm 2: Placebo + Physician's Choice NHA (Placebo Comparator): Placebo + physician's choice NHA (Abiraterone, Darolutamide, or Enzalutamide)
  Interventions: Drug: Placebo; Drug: Abiraterone Acetate; Drug: Darolutamide; Drug: Enzalutamide

INTERVENTIONS:
Drug: Saruparib — Oral
  Other Names: AZD5305
  Arms: Arm 1: Saruparib (AZD5305) + Physician's Choice NHA
Drug: Placebo — Oral
  Arms: Arm 2: Placebo + Physician's Choice NHA
Drug: Abiraterone Acetate — Oral
  Other Names: Zytiga
Drug: Darolutamide — Oral
  Other Names: Nubequa
Drug: Enzalutamide — Oral
  Other Names: Xtandi

SUMMARY:
The intention of the study is to demonstrate superiority of Saruparib (AZD5305) + physician's choice NHA relative to placebo + physician's choice NHA by assessment of radiographic progression-free survival (rPFS) in participants with mCSPC.

DETAILED DESCRIPTION:
Approximately 1800 adult participants with mCSPC will be assigned to one of two cohorts (550 HRRm and 1250 non-HRRm) and randomized in a 1:1 ratio to receive either Saruparib (AZD5305) with NHA or placebo with NHA. They will receive their assigned treatment and regular tumor evaluation scans until disease progression, or until treatment is stopped for another reason.

All patients will be followed for survival until the end of the study. Independent data monitoring committee (DMC) composed of independent experts will be convened to confirm the safety and tolerability of Saruparib (AZD5305) + physicians choice NHA.

ELIGIBILITY:
Inclusion Criteria:

* Male ≥ 18 years of age.
* Histologically documented prostate adenocarcinoma which is de novo or recurrent and castration-sensitive. Participants with pathologic features of small cell, neuroendocrine, sarcomatoid, spindle cell, or signet cell histology are not eligible.
* Metastatic disease as documented by the investigator prior to randomisation, with clear evidence of ≥ 1 bone lesion and/or ≥ 1 soft tissue lesion that is suitable for repeated assessment with CT and/or MRI.
* Participant is receiving ADT with a GnRH analogue or has undergone bilateral orchiectomy starting ≥ 14 days and < 4 months prior to randomisation.
* ECOG performance status of 0 or 1 with no deterioration over the 2 weeks prior to randomisation.
* Provision of FFPE tumour tissue sample and blood sample (for ctDNA).
* Confirmed HRRm status by central tumour tissue and/or ctDNA test is required to determine cohort eligibility.
* Adequate organ and bone marrow function as described in study protocol.
* Participants must not father children or donate sperm from signing ICF, during the study intervention and for 6 months after the last dose of study intervention.
* Participants must use a condom from signing ICF, during study intervention, and for 6 months after the last dose of study drug, with all sexual partners.

Exclusion Criteria:

* Participants with a history of MDS/AML or with features suggestive of MDS/AML (as determined by prior diagnostic investigation). In case there is no clinical MDS/AML suspicion, no specific screening for MDS/AML (by BM/bone biopsy) is required.
* Participants with any known predisposition to bleeding.
* Any history of persisting (> 2 weeks) severe cytopenia.
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD5305 and/or the assigned NHA.
* History of another primary malignancy, with exceptions.
* Persistent toxicities (CTCAE Grade ≥ 2) caused by previous anticancer therapy.
* Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 4 weeks prior to start of study intervention.
* Cardiac criteria, including history of arrhythmia and cardiovascular disease.
* Any prior anticancer pharmacotherapy or surgery for metastatic prostate cancer, with exceptions.
* Prior treatment within 14 days with blood product support or growth factor support.
* Participants who are unevaluable for both bone and soft tissue progression.

Ages: 18 Years to 130 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants
Enrollment: 1800 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2028-01-11 (Estimated); Study Completion 2031-04-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-Free Survival (rPFS) | up to approximately 50 months
  rPFS is defined as the time from randomisation to radiographic progression, as assessed by the investigator per RECIST 1.1 (soft tissue) and/or PCWG3 criteria (bone), or, death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to approximately 90 months
  OS is defined as the time from randomisation until the date of death due to any cause.
Second Progression-Free Survival (PFS2) | up to approximately 50 months
  Time from randomisation to PFS2 is defined as the time from randomisation to the earliest of progression (defined as radiographic progression, clinical progression, or PSA progression) after initiation of first subsequent treatment following the initial investigator-assessed progression or death.
Time to First Subsequent Therapy or Death (TFST) | up to approximately 50 months
  TFST is defined as the time from randomisation to the start date of the first subsequent anticancer therapy after discontinuation of randomised treatment, or death due to any cause.
Symptomatic Skeletal Event-Free Survival (SSE-FS) | up to approximately 50 months
  SSE-FS is defined as the time from randomisation to the earliest of the following:
  * Use of radiation therapy to prevent or relieve skeletal symptoms.
  * Occurrence of new symptomatic pathological bone fractures (vertebral or non-vertebral).
  * Occurrence of spinal cord compression.
  * Orthopaedic surgical intervention for bone metastasis.
  * Death due to any cause.
Time to the First Castration-Resistant Event (TTCR) | up to approximately 50 months
  TTCR is defined as the time from randomisation to the first castration resistant event (radiographic disease progression per RECIST 1.1 [soft tissue] and/or PCWG3 criteria [bone], PSA progression per PCWG3, or SSE, PSA progression per PCWG3, or SSE), whichever occurs first, with castrate levels of testosterone (below 50 ng/dL).
Time to Pain Progression (TTPP) | up to approximately 50 months
  TTPP is defined as the time from randomisation to clinically meaningful pain progression based on a 2-point increase from baseline in the Brief Pain Inventory - Short Form (BPI-SF) Item 3 'worst pain in 24 hours' score and/or initiation of/increase in opioid analgesic use.
Time To Deterioration in Urinary Symptoms (TTDUS) | up to approximately 50 months
  TTDUS is defined as the time from randomisation to deterioration in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Prostate Questionnaire (Urinary Symptoms) (QLQPR25 [US]) subscale scores.
Time to Deterioration in Fatigue (TTDF) | up to approximately 50 months
  TTDF is defined as the time from randomisation to deterioration in Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 7A scores.
Time to Deterioration in Physical Function (TTDPF) | up to approximately 50 months
  TTDPF is defined as the time from randomisation to deterioration in PROMIS Physical Function Short Form 8C scores.
Health-related Quality of Life (HrQoL) | up to approximately 50 months
  Change from baseline in BPI-SF worst pain score, pain severity, and interference domain scores.
BRCA and other HRR gene mutation status. | at screening
Plasma concentrations of AZD5305 | up to approximately 10 months
Samples will be used to develop complementary or companion diagnostics by analyzing their performance characteristics and calculate their consistency with clinical trial assays used for enrolment onto the study. | up to approximately 50 months
  Samples will be tested by a CDx to certify consistency with assays used in the study.
Assessment of PSA (prostate-specific antigen) in participants in mCSPC | up to approximately 50 months
  proportion of participants achieving a >= 50% or >=90% decrease in PSA from baseline; proportion of participants with undetectable PSA (< 0.2 ng/mL); time to PSA progression

OTHER OUTCOMES:
Number of TEAEs (treatment emergent adverse events), SAEs (serious adverse events), and AEs (adverse events) leading to dose modifications | up to approximately 50 months

CONTACTS AND LOCATIONS:
Overall Officials: Kim Nguyen Chi, MD, Principal Investigator — BC Cancer, Canada; Arun Azad, MD, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (344):
- United States (101):
  - Research Site, Chandler, Arizona
  - Research Site, Gilbert, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Springdale, Arkansas
  - Research Site, Bakersfield, California
  - Research Site, Fountain Valley, California
  - Research Site, Fullerton, California
  - Research Site, Los Angeles, California
  - Research Site, Montebello, California
  - Research Site, Pasadena, California
  - Research Site, Pomona, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Barbara, California
  - Research Site, Santa Monica, California
  - Research Site, Santa Rosa, California
  - Research Site, Golden, Colorado
  - Research Site, Lakewood, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Norwich, Connecticut
  - Research Site, Newark, Delaware
  - Research Site, Jacksonville, Florida
  - Research Site, Palm Bay, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Glenview, Illinois
  - Research Site, Lake Barrington, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Westwood, Kansas
  - Research Site, Wichita, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Shreveport, Louisiana
  - Research Site, Scarborough, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Towson, Maryland
  - Research Site, Upper Marlboro, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Billings, Montana
  - Research Site, Bozeman, Montana
  - Research Site, Las Vegas, Nevada
  - Research Site, Belleville, New Jersey
  - Research Site, Brick, New Jersey
  - Research Site, Camden, New Jersey
  - Research Site, East Brunswick, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Rio Rancho, New Mexico
  - Research Site, Albany, New York
  - Research Site, East Syracuse, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Shirley, New York
  - Research Site, Syracuse, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Independence, Ohio
  - Research Site, Wooster, Ohio
  - Research Site, Florence, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Bala-Cynwyd, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Germantown, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Denton, Texas
  - Research Site, Flower Mound, Texas
  - Research Site, Grapevine, Texas
  - Research Site, Houston, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Tyler, Texas
  - Research Site, Wichita Falls, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, St. George, Utah
  - Research Site, Fairfax, Virginia
  - Research Site, Winchester, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Spokane Valley, Washington
  - Research Site, Tacoma, Washington
- Australia (7):
  - Research Site, Chermside
  - Research Site, Darlinghurst
  - Research Site, Hyde Park
  - Research Site, Kurralta Park
  - Research Site, Melbourne
  - Research Site, Randwick
  - Research Site, South Brisbane
- Austria (5):
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Krems
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (4):
  - Research Site, Charleroi
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Leuven
- Brazil (7):
  - Research Site, Curitiba
  - Research Site, Pelotas
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Luís
  - Research Site, São Paulo
- Canada (18):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Abbotsford, British Columbia
  - Research Site, Kelowna, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Halifax, Nova Scotia
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Chile (5):
  - Research Site, Concepción
  - Research Site, La Serena
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (29):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Dongguan
  - Research Site, Guangzhou
  - Research Site, Guilin
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jiaxing
  - Research Site, Jinan
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nantong
  - Research Site, Ningbo
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suining
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Weifang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yantai
  - Research Site, Zhengzhou
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Tampere
  - Research Site, Turku
- France (18):
  - Research Site, Angers
  - Research Site, Bayonne
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nice
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Quimper
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Tours
  - Research Site, Vandœuvre-lès-Nancy
- Germany (29):
  - Research Site, Bergisch Gladbach
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Braunschweig
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Erlangen
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Göttingen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Herne
  - Research Site, Homburg
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, Mettmann
  - Research Site, München
  - Research Site, Münster
  - Research Site, Nürtingen
  - Research Site, Oldenburg
  - Research Site, Regensburg
  - Research Site, Stuttgart
  - Research Site, Trier
  - Research Site, Tübingen
  - Research Site, Ulm
- Hungary (7):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szeged
  - Research Site, Szekszárd
- India (14):
  - Research Site, Bangalore
  - Research Site, Calicut
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Kanpur
  - Research Site, Kolkata
  - Research Site, Mohali
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Surat
  - Research Site, Vadodara
  - Research Site, Varanasi
- Italy (10):
  - Research Site, Bari
  - Research Site, Genoa
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Rome
  - Research Site, Rozzano
  - Research Site, Terni
  - Research Site, Trento
- Japan (26):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Hirakata-shi
  - Research Site, Hirosaki-shi
  - Research Site, Kanazawa
  - Research Site, Kashihara-shi
  - Research Site, Kawagoe-shi
  - Research Site, Kisarazu-shi
  - Research Site, Kita-gun
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sakura-shi
  - Research Site, Sapporo
  - Research Site, Shiwa-gun
  - Research Site, Suita-shi
  - Research Site, Tsu
  - Research Site, Yokohama
  - Research Site, Yufu-shi
- Malaysia (5):
  - Research Site, George Town
  - Research Site, Johor Bahru
  - Research Site, Kota Kinabalu
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Hilversum
  - Research Site, Nijmegen
- Peru (3):
  - Research Site, Arequipa
  - Research Site, Bellavista
  - Research Site, Lima
- Poland (8):
  - Research Site, Bydgoszcz
  - Research Site, Koszalin
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Żory
- Research Site, San Juan, Puerto Rico
- South Korea (4):
  - Research Site, Daejeon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Sabadell
  - Research Site, Valencia
- Sweden (4):
  - Research Site, Gothenburg
  - Research Site, Malmo
  - Research Site, Solna
  - Research Site, Stockholm
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taoyuan District
  - Research Site, Yung Kang City
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khlong Luang
  - Research Site, Songkhla
- Turkey (Türkiye) (5):
  - Research Site, Ankara
  - Research Site, Bornova-Izmir
  - Research Site, Fatih-Istanbul
  - Research Site, Istanbul
  - Research Site, Karşıyaka
- United Kingdom (13):
  - Research Site, Aberdeen
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Glasgow
  - Research Site, Guildford
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne
  - Research Site, Oxford
  - Research Site, Plymouth
  - Research Site, Preston
  - Research Site, Swansea
  - Research Site, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home